CLINICAL TRIAL: NCT01027754
Title: Smoking Cessation Treatment for Methadone Maintenance Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2008-537; UL1RR025750 (NIH)
Record Dates: First submitted 2009-12-07; First posted 2009-12-09 (Estimated); Results first posted 2020-01-29 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Smoking Cessation; Substance-Related Disorders
Keywords: methadone maintenance
MeSH Terms: conditions — Smoking Cessation; Substance-Related Disorders | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Varenicline (Experimental): Drug treatment in combination with telephone quitline referral and brief individual counseling based on PHS guidelines at weeks 2, 4, 8, and 12
  Interventions: Drug: Varenicline
- Placebo (Placebo Comparator): Matched placebo capsules in combination with telephone quitline referral and brief individual counseling based on PHS guidelines at weeks 2, 4, 8, and 12
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Varenicline — Days 1-3: 0.5 mg once a day Days 4-7: 0.5 mg twice a day Days 8-84: 1 mg twice a day
  Other Names: Chantix
  Arms: Varenicline
Drug: Placebo — Days 1-3: 1 pill daily Days 4-7: 2 pills daily Days 8-84: 2 pills daily
  Other Names: Matched capsules
  Arms: Placebo

SUMMARY:
Patients in substance abuse treatment smoke four times more than non-substance abusers, and suffer high rates of tobacco-related disease and death. While many quit smoking treatments exist that have been shown to help non-substance abusers quit smoking, little is known about what treatments work for patients in substance abuse treatment. The drug varenicline (Chantix) has been shown to be more effective at helping people quit smoking than nicotine replacement therapy, bupropion or placebo. However, varenicline has not yet been studied in patients in substance abuse treatment. The study aims to evaluate the feasibility, effectiveness and safety of varenicline, in combination with counseling, in methadone maintained smokers. It also aims to evaluate the link between quitting smoking and alcohol and illicit drug use in methadone maintained smokers. We hypothesize that participants receiving varenicline will have higher abstinence from smoking than participants receiving placebo and that participants taking varenicline will not have significantly more adverse reactions than were described in the general population in other studies. We also hypothesize that compared to continued smokers, tobacco abstainers will be more likely to be abstinent from alcohol or illicit drugs.

DETAILED DESCRIPTION:
Patients in substance abuse treatment smoke four times more than non-substance abusers, and suffer high rates of tobacco-related disease and death. While many quit smoking treatments exist that have been shown to help non-substance abusers quit smoking, little is known about what treatments work for patients in substance abuse treatment. The drug varenicline (Chantix) has been shown to be more effective at helping people quit smoking than nicotine replacement therapy, bupropion or placebo. However, varenicline has not yet been studied in patients in substance abuse treatment. The study aims to evaluate the feasibility, effectiveness and safety of varenicline, in combination with counseling, in methadone maintained smokers. It also aims to evaluate the link between quitting smoking and alcohol and illicit drug use in methadone maintained smokers. We hypothesize that participants receiving varenicline will have higher abstinence from smoking than participants receiving placebo and that participants taking varenicline will not have significantly more adverse reactions than were described in the general population in other studies. We also hypothesize that compared to continued smokers, tobacco abstainers will be more likely to be abstinent from alcohol or illicit drugs.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* English speaking
* Smoked at least 100 cigarettes/lifetime
* Smokes 5 or more cigarettes per day
* Interested in quitting smoking (preparation or contemplation state of change)
* Enrolled in Einstein/Montefiore methadone program for 3 or more months
* Stable methadone dose for 2 weeks
* Agree to use contraception throughout the trial (among women with reproductive potential)
* Willing to participate in all study components
* Able to provide informed consent

Exclusion Criteria:

* Serious or unstable HIV/AIDS, liver, cardiovascular, or pulmonary disease
* Psychiatric instability
* Women who are pregnant, breastfeeding, or contemplating pregnancy
* Creatinine clearance less than 30 mL/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2009-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shadi Nahvi, M.D., M.S., Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine of Yeshiva University, The Bronx, New York, United States

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- [Derived] Nahvi S, Ning Y, Segal KS, Richter KP, Arnsten JH. Varenicline efficacy and safety among methadone maintained smokers: a randomized placebo-controlled trial. Addiction. 2014 Sep;109(9):1554-63. doi: 10.1111/add.12631. Epub 2014 Jun 27. PMID 24862167

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Varenicline | Placebo
Started | 57 | 55
Completed | 55 | 47
Not Completed | 2 | 8
Not completed — withdrew/lost to follow-up after interve | 2 | 3
Not completed — Withdrawal by Subject | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline | Placebo | Total
Number analyzed (Participants) | 57 | 55 | 112
Age, Customized [Mean (Standard Deviation); unit: years]
  Age, Customized | 48 (9) | 48 (8) | 48 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 28 | 59
  Male | 26 | 27 | 53
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic | 32 | 28 | 60
  Black | 14 | 17 | 31
  Non-Hispanic white | 5 | 5 | 10
  Other | 6 | 5 | 11
Less than/equal to high school education, [Number; unit: participants] | 41 | 46 | 87
Married or living with partner [Number; unit: participants] | 23 | 31 | 54
Employed [Number; unit: participants] | 15 | 17 | 32
Life-time history of incarceration [Number; unit: participants] | 42 | 31 | 73
Unstable housing, [Number; unit: participants] | 21 | 14 | 35
Cigarettes/day, median (IQR) [Median (Inter-Quartile Range); unit: cigarettes/day] | 15 [10 to 20] | 15 [10 to 20] | 15 [10 to 20]
Carbon monoxide, median (IQR) [Median (Inter-Quartile Range); unit: p.p.m.] — Population: Carbon monoxide, median (IQR) (n=107). The number analyzed in row differs from overall due to missing data for the carbon monoxide variable because the total n for the paper was 112.
  p.p.m.
    number analyzed (Participants) | 55 | 52 | 107
    (all) | 10 [6 to 15] | 9 [7 to 17] | 10 [6 to 15]
Carbon monoxide < 8 p.p.m., [Number; unit: participants] — Population: The number analyzed in row differs from overall due to missing data for the carbon monoxide variable because the total n for the paper was 112.
  participants
    number analyzed (Participants) | 55 | 52 | 107
    (all) | 22 | 18 | 40
Fagerström Test of Nicotine Dependence score, median (IQR) [Median (Inter-Quartile Range); unit: units on a scale] — 6 item scale, with scores ranging from 0 - 10 score under 3 = low nicotine dependence, 4-5 = moderate nicotine dependence, and 6-10 = high nicotine dependence
  units on a scale | 4 [2 to 6] | 4 [3 to 5] | 4 [2 to 5]
Ladder of change score, median (IQR) [Median (Inter-Quartile Range); unit: units on a scale] — Ladder of Change is to assess a smoker's position on a continuum (scale of 1 to 10) ranging from having no thoughts of quitting (1) to having quit smoking (10).
  units on a scale | 7 [6 to 8] | 7 [6 to 8] | 7 [6 to 8]
Quit importance, median (IQR) [Median (Inter-Quartile Range); unit: units on a scale] — Importance of quitting smoking measured on a scale of 1-10 (10 = high levels of quit importance).
  units on a scale | 10 [8 to 10] | 10 [9 to 10] | 10 [8 to 10]
Quit confidence, median (IQR) [Median (Inter-Quartile Range); unit: units on a scale] — Confidence of quitting smoking measured on a scale of 1-10 (10 = high levels of quit confidence).
  units on a scale | 8 [5 to 9] | 8 [5 to 10] | 8 [5 to 10]
Any past quit attempts, n [Number; unit: participants] | 41 | 41 | 82
Median duration longest prior quit attempt, weeks (IQR) [Median (Inter-Quartile Range); unit: weeks] — Population: n=82 participants who reported any past quit attempts queried
  weeks
    number analyzed (Participants) | 41 | 41 | 82
    (all) | 9 [1 to 30] | 4 [1 to 26] | 4.3 [1 to 30]
Any other household smoker [Number; unit: participants] | 34 | 29 | 63
Life-time major depressive disorder [Number; unit: participants] | 12 | 11 | 23
Life-time psychotic disorder, n [Number; unit: participants] | 9 | 9 | 18
Life-time suicide attempt, n [Number; unit: participants] | 9 | 7 | 16
Severe global psychiatric symptoms, n [Number; unit: participants] | 9 | 12 | 21
Currently receiving psychiatric treatment, n [Number; unit: participants] | 24 | 26 | 50
Hypertension, n [Number; unit: participants] | 19 | 22 | 41
Diabetes, n [Number; unit: participants] | 13 | 11 | 24
COPD/asthma, n [Number; unit: participants] | 19 | 12 | 31
HIV/AIDS, n [Number; unit: participants] | 11 | 10 | 21
Median duration methadone maintenance, years (IQR) [Median (Inter-Quartile Range); unit: years] | 4 [2 to 10] | 7 [3 to 13] | 5.9 [2.4 to 10.9]
Median methadone dose, mg (IQR) [Median (Inter-Quartile Range); unit: milligram] | 110 [70 to 150] | 100 [65 to 160] | 110 [70 to 160]
Self reported use of heroin in 30 days prior to baseline, n [Number; unit: participants] | 8 | 5 | 13
Self reported use of other opiates in 30 days prior to baseline, n [Number; unit: participants] | 11 | 13 | 24
Self reported use of cocaine (including crack) in 30 days prior to baseline, n [Number; unit: participants] | 17 | 8 | 25
Self reported use of marijuana in 30 days prior to baseline, n [Number; unit: participants] | 14 | 13 | 27
Self reported use of hazardous alcohol use in 30 days prior to baseline, n [Number; unit: participants] | 4 | 9 | 13
Participants enrolled at clinical site 1, n [Number; unit: participants] | 9 | 7 | 16
Participants enrolled at clinical site 2, n [Number; unit: participants] | 32 | 33 | 65
Participants enrolled at clinical site 3, n [Number; unit: participants] | 16 | 15 | 31

OUTCOME MEASURES:

1. Primary Outcome: Biochemically Verified Abstinence Verified With Expired Carbon Monoxide (CO) < 8 p.p.m.
Time Frame: Week 12
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 57 | 55
participants | 6 | 0
Statistical Analysis 1: Comparison: Varenicline vs Placebo; Test type: Superiority or Other; p = 0.03, Fisher Exact

2. Secondary Outcome: Biochemically Verified Abstinence Verified With Expired Carbon Monoxide (CO) < 8 p.p.m.
Time Frame: Week 24
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 57 | 55
participants | 3 | 0
Statistical Analysis 1: Comparison: Varenicline vs Placebo; Test type: Superiority or Other; p = 0.24, Fisher Exact

3. Secondary Outcome: Number of Counseling Visits Completed
Description: Participants were offered 5 counseling visits at weeks 0, 2, 4, 8, 12.
Time Frame: End of 12 week intervention period
Measure: Mean (Standard Deviation); unit: visits completed
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 57 | 55
visits completed | 1.96 (1.64) | 1.85 (1.65)

4. Secondary Outcome: Number of Study Visits Completed
Description: Mean number of study visit completed out of a possible total of 6 study visits at weeks 0, 2, 4, 8, 12 and 24.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: visits completed
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 57 | 55
visits completed | 5.72 (0.70) | 5.36 (1.38)

5. Secondary Outcome: 7-day Point Prevalence Abstinence at 12 Weeks as Verified by Salivary Cotinine.
Description: Threshold of salivary cotinine ≤ 15 ng/ml was prespecified. Salivary cotinine was measured among participants who self-reported 7-day point prevalence abstinence using a semi-quantitative assay (Nymox NicAlert™).
Time Frame: Weeks 2, 4, 8, 12, and 24
Population: Because of the high rate of missing data (6 of 51 cases of self-reported abstinence not verified by cotinine), and because the semi-quantitative assay we used (Nymox NicAlert™) did not use a ≤ 15 ng/ml threshold (10 of 51 cases fell in the 10-30 ng/ml range), this data was not analyzed.
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Cigarettes Smoked Per Day
Time Frame: Weeks 2, 4, 8, 12, and 24
Measure: Median (Inter-Quartile Range); unit: cigarettes/day
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 57 | 55
cigarettes/day
  At week 2 | 3 [1 to 9] | 6 [3 to 10]
  At week 4 | 2 [0.5 to 7] | 5 [3 to 10]
  At week 8 | 3 [1 to 6] | 5 [3 to 10]
  At week 12 | 2 [0.5 to 2] | 5 [2 to 10]
  At week 24 | 4 [2 to 7] | 5 [2.5 to 10]

7. Secondary Outcome: Number of Participants With an Attempt to Quit Smoking That Lasted ≥ 24 Hours
Time Frame: Weeks 2, 4, 8, 12, and 24
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 57 | 55
participants
  At week 2 | 33 | 25
  At week 4 | 35 | 27
  At week 8 | 37 | 32
  At week 12 | 37 | 25
  At week 24 | 41 | 30

8. Secondary Outcome: Confidence in Quitting Smoking (1-10 Scale)
Description: Confidence of quitting smoking measure on a scale of 1-10 (10= high levels of quit confidence).
Time Frame: Weeks 2, 4, 8, 12, and 24
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 57 | 55
units on a scale
  At week 2 | 8 [7 to 10] | 8 [6 to 10]
  At week 4 | 9 [6 to 10] | 8 [7 to 10]
  At week 8 | 9 [7 to 10] | 9 [7 to 10]
  At week 12 | 9 [7 to 10] | 8 [6 to 10]
  At week 24 | 8 [6 to 10] | 8 [5 to 10]

9. Secondary Outcome: Importance of Quitting Smoking (1-10 Scale)
Description: Importance of quitting smoking measured on a scale of 1-10 (10=high levels of quit importance).
Time Frame: Weeks 2, 4, 8, 12, and 24
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 57 | 55
units on a scale
  At week 2 | 10 [10 to 10] | 10 [9 to 10]
  At week 4 | 10 [10 to 10] | 10 [9 to 10]
  At week 8 | 10 [10 to 10] | 10 [9 to 10]
  At week 12 | 10 [10 to 10] | 10 [9 to 10]
  At week 24 | 10 [10 to 10] | 10 [8 to 10]

10. Secondary Outcome: Adverse Medication Effects
Time Frame: over the intervention period (measured at weeks 2, 4, 8, 12, and 24)
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 57 | 55
participants
  Change in taste | 18 | 14
  Dry Mouth | 27 | 23
  Change in appetite | 29 | 18
  Nausea | 29 | 14
  Vomiting | 11 | 8
  Gas | 19 | 15
  Constipation | 23 | 9
  Change in concentration | 6 | 6
  Headache | 11 | 18
  Fatigue | 15 | 13
  Insomnia | 15 | 13
  Dizziness | 9 | 8
  Irritability | 10 | 8
  Vivid/more frequent dreams | 18 | 22

11. Secondary Outcome: Number of Participants With Severe Global Psychiatric Symptoms Assessed by the Brief Symptom Inventory
Time Frame: over the intervention period (measured at weeks 2, 4, 8, 12, and 24)
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 57 | 55
participants
  Week 2 | 9 | 11
  Week 4 | 4 | 7
  Week 8 | 6 | 7
  Week 12 | 8 | 5
  Week 24 | 5 | 5
Statistical Analysis 1: Comparison: Varenicline vs Placebo; Test type: Superiority or Other; p = 0.15, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Number of Patients With Suicial Ideation (Wishes to be Dead, or Thoughts of Killing Self) Assessed Using the Columbia Suicide Severity Scale
Time Frame: over the intervention period (measured at weeks 2, 4, 8, 12, and 24)
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 57 | 55
participants
  Week 2 | 1 | 1
  Week 4 | 1 | 0
  Week 8 | 1 | 1
  Week 12 | 1 | 2
  Week 24 | 1 | 1

13. Secondary Outcome: Number of Participants With Major Depressive Episode, Assessed by the Mini-International Neuropsychiatric Interview
Time Frame: over the intervention period (measured at weeks 2, 4, 8, 12, and 24)
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 57 | 55
participants
  Week 2 | 0 | 0
  Week 4 | 0 | 0
  Week 8 | 2 | 0
  Week 12 | 0 | 1
  Week 24 | 2 | 2

14. Secondary Outcome: Number of Participants With Manic Episode, Assessed by the Mini-International Neuropsychiatric Interview
Time Frame: over the intervention period (measured at weeks 2, 4, 8, 12, and 24)
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 57 | 55
participants
  Week 2 | 0 | 0
  Week 4 | 0 | 0
  Week 8 | 0 | 0
  Week 12 | 0 | 0
  Week 24 | 0 | 0

15. Secondary Outcome: Number of Participants With Psychotic Disorder, Assessed by the Mini-International Neuropsychiatric Interview
Time Frame: over the intervention period (measured at weeks 2, 4, 8, 12, and 24)
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 57 | 55
participants
  Week 2 | 0 | 2
  Week 4 | 0 | 0
  Week 8 | 1 | 0
  Week 12 | 1 | 1
  Week 24 | 2 | 1

ADVERSE EVENTS:
Description: Adverse events were assess using both a structured questionnaire that assessed the presence of specific symptoms reported among varenicline subjects in published clinical trials, and an open-ended review of symptoms that emerged or increased in intensity following the start of study medication. Serious adverse events were defined as those which resulted in death, were life-threatening or required in-patient hospitalization.
Arm/Group | Varenicline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/55
Serious Adverse Events (participants affected / at risk) | 3/57 | 2/55
Other Adverse Events (participants affected / at risk) | 52/57 | 46/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline (N=57) | Placebo (N=55)
Hypoglycemic episode preceding increase in long-acting insulin dose (Endocrine disorders) | 1 | 0
Hospitalization for alcohol and cocaine rehabilitation (Endocrine disorders) | 1 | 0
Knee replacement following mechanical fall (Musculoskeletal and connective tissue disorders) | 1 | 0
Hospitalization for chest pain (Cardiac disorders) | 0 | 1
Hospitalization for alcohol detoxification (Endocrine disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline (N=57) | Placebo (N=55)
Psychiatric outcome: incident major depressive episode (Psychiatric disorders) | 2 | 1
Psychiatric outcome: incident manic episode (Psychiatric disorders) | 0 | 0
Psychiatric outcome: Incident psychotic disorder (Psychiatric disorders) | 1 | 3
Psychiatric outcome: suicidal ideation (Psychiatric disorders) | 3 | 4
Psychiatric outcome: severe global psychiatric symptoms (Psychiatric disorders) | 12 | 17
Medical symptom: change in taste (Respiratory, thoracic and mediastinal disorders) | 18 | 14
medical symptom: dry mouth (General disorders) | 27 | 23
medical symptom: change in appetite (Metabolism and nutrition disorders) | 29 | 18
medical symptom: nausea (Gastrointestinal disorders) | 29 | 14
medical symptom: vomiting (Gastrointestinal disorders) | 11 | 8
medical symptom: gas (Gastrointestinal disorders) | 19 | 15
medical symptom: constipation (Gastrointestinal disorders) | 23 | 9
medical symptom: change in concentration (Nervous system disorders) | 6 | 6
Medical Symptom: headache (Nervous system disorders) | 11 | 18
medical symptom: fatigue (General disorders) | 15 | 13
medical symptom: insomnia (Psychiatric disorders) | 15 | 13
medical symptom: dizziness (General disorders) | 9 | 8
medical symptom: irritability (Nervous system disorders) | 10 | 8
medical symptom: vivid/more frequent dreams (Nervous system disorders) | 18 | 22

LIMITATIONS AND CAVEATS:
Self-reported smoking reduction could not be biochemically validated. We did not analyze changes in drug use over time. Sample size limited power to detect rare psychiatric events. Findings may not be generalizable to other populations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No